CLINICAL TRIAL: NCT05964829
Title: A Crossover Study Evaluating the Impact of the Cionic Neural Sleeve on Mobility, Disability, Fall Risk, and Physical Activity in Multiple Sclerosis
Brief Title: Impact of the Cionic Neural Sleeve on Mobility in Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cionic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CIONIC-06-001
Record Dates: First submitted 2023-07-18; First posted 2023-07-28 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Experimental): Participants will follow the walking program.
  Interventions: Behavioral: Walking Program
- Functional electrical stimulation (Experimental): Participants will follow the walking program and receive stimulation assistance during the walking sessions.
  Interventions: Device: Cionic Neural Sleeve NS-100; Behavioral: Walking Program

INTERVENTIONS:
Device: Cionic Neural Sleeve NS-100 — The Cionic Neural Sleeve applies functional electrical stimulation as subjects walk to help contract appropriate muscles at appropriate times. The Cionic Neural Sleeve will be worn for 6 weeks.
  Arms: Functional electrical stimulation
Behavioral: Walking Program — 15 minutes of walking for 5 days per week for 6 weeks

SUMMARY:
The purpose of this research is to support the clinical value of the Cionic Neural Sleeve for individuals diagnosed with multiple sclerosis (MS).

DETAILED DESCRIPTION:
The randomized within-participants crossover 12-week study aims to demonstrate the clinical impact of the Cionic Neural Sleeve for individuals diagnosed with MS.

Physical measurements, performance-based tests, and questionnaire responses will be recorded. These include physical activity recorded by the Cionic Neural Sleeve; in-person tests measuring disability, spasticity and balance; and questionnaires gauging perceived walking ability, quality of life, and physical and psychological impact of MS.

All participants will be assigned a Cionic Neural Sleeve on the most impacted leg for 6 weeks, and prescribed a home-based intervention of 15 minutes of walking for 5 days a week for 12 weeks. The Cionic Neural Sleeve will be worn for 6 weeks of the study while following the walking program.

Participants will be randomized to one of two groups: A or B. Group A will follow the walking program and wear the Neural Sleeve to receive stimulation assisted walking from the Neural Sleeve for 6 weeks. Group B will follow the walking program for 6 weeks. After 6 weeks, participants in each group will cross over to the other group.

ELIGIBILITY:
Inclusion Criteria:

* Persons with relapsing-remitting or progressive forms of MS between the ages of 22 and 75
* Ability to ambulate at least 15 minutes throughout the day for five days per week, with or without assistive device
* Adequate cognitive and communicative function as assessed via Telephone Interview for Cognitive Status (TICS) to identify persons with dementia
* Able to tolerate the Neural Sleeve device for up to 8 hours per day
* T25FWT time between 8 and 45 seconds
* No recent change in medication or recent exacerbation of symptoms over the last 60 days
* Patient-determined Disease Steps score between 3 and 5 or EDSS score between 4 and 6.5

Exclusion Criteria:

* Lower motor neuron disease or injury (e.g. peripheral neuropathy) that may impair response to stimulation
* Absent sensation in the impacted or more impacted leg
* Inadequate response to stimulation, defined by inability to achieve muscle contraction or unable to tolerate stimulation
* Inability to ambulate with the sleeve in place of an ankle foot orthosis (AFO)/knee ankle foot orthosis (KAFO) if utilized
* History of falls greater than once a week
* No use of FES devices in the past year
* Demand-type cardiac pacemaker or defibrillator
* Malignant tumor in the impacted or more impacted leg
* Existing thrombosis in the impacted or more impacted leg
* Fracture or dislocation in the impacted or more impacted leg that could be adversely affected by motion from stimulation

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Gait Speed | Day 0, Week 6, Week 12
  The Timed 25-Foot Walk Test (T25FWT) to record duration of time to walk a distance of 25 feet, measured in seconds. The score is the average of two successive trials.
Change in Perceived Walking Ability | Day 0, Week 6, Week 12
  Multiple Sclerosis Walking Scale-12 (MSWS-12) to measure perceived impact of MS on walking ability, measured by score. Scores on the MSWS-12 range from 12-60 and transformed to a scale with a range from 0 to 100, with high scores indicative of a greater impact of MS on walking.
Change in MS Disability | Day 0, Week 6, Week 12
  A 9-item survey, Patient-Determined Disease Steps (PDDS), will measure of disability status in individuals with MS. The PDDS ranges from 0 to 8, with higher values indicative of higher levels of disability.
Amount of Daily Walking/Activity Level | During allocation to receive the functional electrical stimulation arm
  Collected by the usage log of the device, measured in steps per day
Duration of Daily Walking/Activity Level | During allocation to receive the functional electrical stimulation arm
  Collected by the usage log of the device, measured in duration of activity.

OTHER OUTCOMES:
Change in Health-Related Quality of Life | Day 0, Week 6, Week 12
  The Euroqol 5 Dimension 5 Level (EQ-5D-5L) questionnaire describes health profiles using different domains, measured by a 5-digit code. Single-digit numbers of the dimensions range from 1 to 5, with 1 indicative of no problem and 5 indicative of extreme problems in that domain.
Change in Impact of MS | Day 0, Week 6, Week 12
  Multiple Sclerosis Impact Scale-29 (MSIS-29) questionnaire to measure the physical and psychological impact of MS, measured by score. Scores on the MSIS-29 are transformed into a score out of 100, with higher scores indicative of greater degree of disability.
Change in Perceived Fatigue | Day 0, Week 6, Week 12
  Modified Fatigue Impact Scale (MFIS) survey to measure the effects of fatigue in physical, cognitive, and psychosocial functioning. MFIS score ranges from 0 to 84, with high scores indicative of a greater impact of fatigue on activities.
Change in Spasticity | Day 0, Week 6, Week 12
  A trained clinician will administer the Modified Ashworth Scale (MAS) to assess for muscle tone and spasticity. Scores of the MAS range from 0 to 4, with high scores representative of increased muscle tone and spasticity.
Change in Lower Limb Strength | Day 0, Week 6, Week 12
  Strength assessment of the ankle dorsiflexors, hamstrings, and quadriceps muscles using a handheld dynamometer in seated or laying in prone, measured in Newtons.
Change in Ankle Plantarflexor Strength | Day 0, Week 6, Week 12
  Ankle plantarflexor strength will be measured by maximal repetitions of single leg heel raises.
Change in Lower Limb Range of Motion | Day 0, Week 6, Week 12
  Range of motion of the ankle, knee, and hips will be assessed by a trained clinician using a handheld goniometer.
Change in Walking Endurance | Day 0, Week 6, Week 12
  Measured via the 6-minute walk test, where subjects will walk as far as possible for 6 minutes, measured in meters.
Change in Balance | Day 0, Week 6, Week 12
  Measured using force platform posturography in standing to quantify postural sway. There will be four 30-second trials with eyes open standing as still as possible.
Change in Incidence of Falls | From enrollment to end of treatment at 12 weeks
  Measured using a self-reported fall diary and a survey, the Hopkins Fall Grading Scale, a 4-point scale to grade the nature and severity of a fall. Higher grades represent increased severity and impact of injurious falls.
Change in Medication(s) and Dosage | Day 0, Week 6, Week 12
  Measured by changes in dose intensities of prescribed medication(s).
Change in Pain | Day 0, Week 6, Week 12
  Measured using the questionnaire, the Numeric Pain Rating Scale (NPRS), an 11-point numeric scale ranging from 0 to 10, with 0 being no pain and 10 being worst pain imaginable.
Change in Self-Reported Physical Activity | From enrollment to end of treatment at 12 weeks
  Subjects will record their weekly physical activity using the Godin-Leisure Time Exercise Questionnaire (GLTEQ), measured by score. Scores less than 14 units are interpreted as insufficiently active/sedentary, while scores between 14 and 23 are interpreted as moderately active, and scores greater than 24 units are interpreted as active.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas A Wajda, PhD, Principal Investigator — Cleveland State University
Locations (1):
- Cleveland State University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No